CLINICAL TRIAL: NCT05657860
Title: A Double Blind, Placebo Controlled, Fixed-Flexible Dose Clinical Trial of Guanfacine Extended Release for the Reduction of Aggression and Self-injurious Behavior Associated With Prader-Willi Syndrome
Brief Title: Guanfacine Extended Release for the Reduction of Aggression and Self-injurious Behavior Associated With Prader-Willi Syndrome
Acronym: PWS-GXR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2020-11-03-MMC
Record Dates: First submitted 2022-12-12; First posted 2022-12-20 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Prader-Willi Syndrome; Aggression; Self-Injurious Behavior; Pathologic Processes; Behavioral Symptoms; Intellectual Disability; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Abnormalities, Multiple; Congenital Abnormalities; Chromosome Disorders; Genetic Diseases, Inborn; Obesity; Overnutrition; Nutrition Disorders; Antihypertensive Agents; Neurotransmitter Agents; Molecular Mechanisms of Pharmacological Action; Physiological Effects of Drugs; Skin-Picking
Keywords: Adrenergic alpha-2 Receptor Agonist; Guanfacine; Adrenergic alpha-Agonists; Adrenergic Agonists; Adrenergic Agents
MeSH Terms: conditions — Prader-Willi Syndrome; Aggression; Self-Injurious Behavior; Pathologic Processes; Behavioral Symptoms; Intellectual Disability; Neurobehavioral Manifestations; Neurologic Manifestations; Nervous System Diseases; Abnormalities, Multiple; Congenital Abnormalities; Chromosome Disorders; Genetic Diseases, Inborn; Obesity; Overnutrition; Nutrition Disorders; Excoriation Disorder | interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Placebo (Sham Comparator)
  Interventions: Other: Placebo
- GXR (Experimental): Immediately following the 8-week blinded randomized trial, an 8-week open-label continuation phase will be pursued to further define efficacy and tolerability of GXR, and to establish its safety with specific focus on metabolic profile.
  Interventions: Drug: Guanfacine Extended Release

INTERVENTIONS:
Drug: Guanfacine Extended Release — Initial dose for all participants will be 1mg per day. If the medication is well tolerated, the dose can be raised to 2 mg until day 28 and increased to 3 mg for the remaining 4 weeks in the trial. The dose schedule will not be fixed., the treating clinician can delay a planned increase or lower the dose to manage adverse effects. At week 8 timepoint, the study will be unblinded.and subjects will continue treatment for 8 weeks.
  Other Names: Intuniv
  Arms: GXR
Other: Placebo — Placebo will be administered concurrently with GXR during trials.
  Arms: Placebo

SUMMARY:
This is a placebo-controlled clinical trial to assess whether Guanfacine Extended Release (GXR) reduces aggression and self injurious behavior in individuals with Prader Willi Syndrome (PWS). In addition, the study will establish the safety of GXR with a specific focus on metabolic effects.

DETAILED DESCRIPTION:
Prader-Willi syndrome is a genetic disorder due to loss of function of specific genes. In newborns, symptoms include weak muscles, poor feeding, and slow development. Beginning in childhood, the person becomes constantly hungry, which often leads to obesity and type 2 diabetes. Aggression, oppositional behavior, and temper tantrums frequently occur in patients with PWS. PWS also has a high prevalence of self-injury, repetitive behavior, impulsivity, over-activity, and mild to moderate learning disability.

Guanfacine Extended Release (GXR), the investigational drug in this study would be the first study to evaluate the drug in patients with Prader Willi Syndrome. "Investigational" means it is not approved by the Food and Drug Administration (FDA) to treat Prader Willi Syndrome. However, Guanfacine Extended Released (GXR) is an FDA approved drug used to treat children and adolescents with hypertension and attention deficit hyperactivity disorder (ADHD). GXR is thought to respond to parts of the brain that lead to strengthening working memory, reducing distraction, improving attention and impulse control. GXR is generally considered safe for children as long as it is used according to the dosing instructions (up to 4mg) of a qualified medical professional.

This randomized, double-blind, placebo-controlled clinical trial aims to determine whether guanfacine extended release (GXR) reduces aggression and self-injury compared to placebo in individuals with PWS with moderate to severe aggressive and/or self-injurious behavior. In addition, GXR's tolerability will be assessed by systematically evaluating and documenting adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PWS confirmed by genetic testing documentation
* Rating of moderate or above on the Clinical Global Impression- Severity Scale

Exclusion Criteria:

* Subjects with positive pregnancy test, swallowing difficulty, and/or presenting with active psychosis or mania will be excluded
* Subjects currently taking guanfacine extended release
* Patients with lactose intolerance
* Individuals with pre-existing, clinically significant bradycardia (< 8 years: <64 bpm; 8 to 12 years: <59 bpm; 12 to 16 years: <53 bpm) or hypotension, defined as 5th percentile for height and gender,26 will be excluded from the study.
* Subjects receiving antipsychotic medications due to a documented history of psychosis or bipolar disorder will be allowed to continue taking the medication without dosage modification.
* Growth hormone, thyroid hormone replacement treatment, and non-psychiatric medicines will be allowed to continue.
* N-Acetyl Cysteine and anticonvulsant medication (only if prescribed for seizures) will be allowed to continue, with specific instructions to not make any dosage changes during the clinical trial.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-17 (Actual); Primary Completion 2023-12-16 (Actual); Study Completion 2023-12-16 (Actual)

PRIMARY OUTCOMES:
Clinical Global Impression- Improvement change from baseline to week 16 | 16 Weeks
  Clinical Global Impression-Improvement is a 7 item scale. A rating of 0=not assessed, 1= very much improved, 2= much improved, 3=minimally improved, 4= no change, 5= minimally worse, 6= much worse, and 7= very much worse. Scores after "4" indicate a decreasing health outcome. Positive clinical response will be determined by a rating of 1= very much improved or 2= Much improved at the end of the blinded trial.

SECONDARY OUTCOMES:
A change in Aberrant Behavior Checklist from baseline to week 16 | 16 Weeks
  Aberrant Behavior Checklist is a 58 item survey. Items are rated on 4 point scale, "0" indicates no problem, "3" indicates major problem. Higher scores are associated with greater severity. The scales are subdivided into 5 subscales: hyperactivity, lethargy, stereotypical behavior, irritability, and inappropriate speech.
A change in Self-Injury Trauma Scale from baseline to week 16 | 16 Weeks
  Self Injury Trauma Scale is divided into three parts. Part 1 is an observation of healed injuries and identifying self injurious behaviors. Part 2 is subdivided into three parts number, type, and severity. Number is based on the number of wounds 1=one wound (common in a mild cases but rare in a severe case) 2=two or four wounds (common) and 3=five or more wounds (rare). Type is categorical and used to differentiate between abrasion/laceration and contusion. Injury severity is scored on a 3 item scale. "1" represents the least severe option and "3" represents the most severe option. Injury severity is broken down between type. Part 3 is the Estimate of Current Risk. It is assessed on a subjective basis with labels such as "mild", "moderate", and "severe" accompanied by descriptions of the observed state of the anatomy. Higher scores are associated with greater severity.
A change in Modified Overt Aggression Scale from baseline to week 16 | 16 Weeks
  Modified Overt Aggression Scale is a four-part behavior rating scale used to evaluate and document the "frequency and severity" of aggressive episodes. The rating scale is made up of four categories: verbal aggression, aggression against objects, aggression against self, and aggression against others. Each part is rated on a 5 point scale, "0" indicates no aggression, "4" indicates the most aggressive option. Higher scores are associated with greater severity.

CONTACTS AND LOCATIONS:
Overall Officials: Deepan Singh, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daly EJ, Trivedi MH, Janik A, Li H, Zhang Y, Li X, Lane R, Lim P, Duca AR, Hough D, Thase ME, Zajecka J, Winokur A, Divacka I, Fagiolini A, Cubala WJ, Bitter I, Blier P, Shelton RC, Molero P, Manji H, Drevets WC, Singh JB. Efficacy of Esketamine Nasal Spray Plus Oral Antidepressant Treatment for Relapse Prevention in Patients With Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2019 Sep 1;76(9):893-903. doi: 10.1001/jamapsychiatry.2019.1189. PMID 31166571
- [Background] Wajs E, Aluisio L, Holder R, Daly EJ, Lane R, Lim P, George JE, Morrison RL, Sanacora G, Young AH, Kasper S, Sulaiman AH, Li CT, Paik JW, Manji H, Hough D, Grunfeld J, Jeon HJ, Wilkinson ST, Drevets WC, Singh JB. Esketamine Nasal Spray Plus Oral Antidepressant in Patients With Treatment-Resistant Depression: Assessment of Long-Term Safety in a Phase 3, Open-Label Study (SUSTAIN-2). J Clin Psychiatry. 2020 Apr 28;81(3):19m12891. doi: 10.4088/JCP.19m12891. PMID 32316080
- [Background] Ochs-Ross R, Daly EJ, Zhang Y, Lane R, Lim P, Morrison RL, Hough D, Manji H, Drevets WC, Sanacora G, Steffens DC, Adler C, McShane R, Gaillard R, Wilkinson ST, Singh JB. Efficacy and Safety of Esketamine Nasal Spray Plus an Oral Antidepressant in Elderly Patients With Treatment-Resistant Depression-TRANSFORM-3. Am J Geriatr Psychiatry. 2020 Feb;28(2):121-141. doi: 10.1016/j.jagp.2019.10.008. Epub 2019 Oct 17. PMID 31734084
- [Background] Ketterer MW, Brymer J, Rhoads K, Kraft P, Lovallo WR. Is aspirin, as used for antithrombosis, an emotion-modulating agent? J Psychosom Res. 1996 Jan;40(1):53-8. doi: 10.1016/0022-3999(95)00524-2. PMID 8730644
- [Background] Mendlewicz J, Kriwin P, Oswald P, Souery D, Alboni S, Brunello N. Shortened onset of action of antidepressants in major depression using acetylsalicylic acid augmentation: a pilot open-label study. Int Clin Psychopharmacol. 2006 Jul;21(4):227-31. doi: 10.1097/00004850-200607000-00005. PMID 16687994
- [Background] Ng QX, Ramamoorthy K, Loke W, Lee MWL, Yeo WS, Lim DY, Sivalingam V. Clinical Role of Aspirin in Mood Disorders: A Systematic Review. Brain Sci. 2019 Oct 29;9(11):296. doi: 10.3390/brainsci9110296. PMID 31671812
- [Background] Marland S, Ellerton J, Andolfatto G, Strapazzon G, Thomassen O, Brandner B, Weatherall A, Paal P. Ketamine: use in anesthesia. CNS Neurosci Ther. 2013 Jun;19(6):381-9. doi: 10.1111/cns.12072. Epub 2013 Mar 22. PMID 23521979
- [Background] Motov S, Rockoff B, Cohen V, Pushkar I, Likourezos A, McKay C, Soleyman-Zomalan E, Homel P, Terentiev V, Fromm C. Intravenous Subdissociative-Dose Ketamine Versus Morphine for Analgesia in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2015 Sep;66(3):222-229.e1. doi: 10.1016/j.annemergmed.2015.03.004. Epub 2015 Mar 26. PMID 25817884